CLINICAL TRIAL: NCT01748344
Title: A Randomised, Placebo Controlled, Four Period Crossover Study to Evaluate the Efficacy, Safety of Oral Repeat Doses of ONO-4053 and Cetirizine in Subjects With Seasonal Allergic Rhinitis in the Vienna Challenge Chamber.
Brief Title: Phase II Study Evaluating ONO-4053 and Cetirizine in Subjects With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ONO-4053POE003
Record Dates: First submitted 2012-11-01; First posted 2012-12-12 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2012-09

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental 1 (Experimental): High dose ONO-4053
  Interventions: Drug: High dose ONO-4053
- Cetirizine (Active Comparator): 10mg Cetirizine
  Interventions: Drug: Cetirizine
- Experimental 2 (Experimental): Low dose ONO-4053
  Interventions: Drug: Low dose ONO-4053
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cetirizine — 10mg tablets
  Arms: Cetirizine
Drug: High dose ONO-4053 — Experimental
  Other Names: Experimental 1
  Arms: Experimental 1
Drug: Low dose ONO-4053 — Experimental
  Other Names: Experimental 2
  Arms: Experimental 2
Drug: Placebo — None active
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate if ONO-4053 relieves symptoms of allergic rhinitis in seasonal allergic rhinitis subjects exposed to pollen under controlled conditions.

DETAILED DESCRIPTION:
The purpose of this study is to investigate if ONO-4053 will impact allergic rhinitis symptoms in subjects with seasonal allergic rhinitis when they are exposed to pollen administered at a fixed rate in an inhalation exposure chamber compared to the standard treatment Cetirizine 10mg under the same conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged between 18 and 65 years inclusive, and healthy with the exception of allergic rhinitis or mild asthma that does not require treatment and has provided written informed consent, which signifies an agreement to enter the study and comply with the restrictions and requirements listed in the informed consent form.
* The subject exhibits a moderate to severe response to grass pollen grains in the allergen challenge chamber at Screening.

Exclusion Criteria:

* The subject on examination is found to have nasal structural abnormalities or nasal polyps; a history of frequent nose bleeds, nasal biopsy, nasal trauma or nasal surgery.
* Pregnant or breast-feeding females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score | 4 months
  To investigate the effect of repeat oral doses of ONO-4053 versus placebo on nasal symptoms elicited by allergen chamber challenge in subjects with seasonal allergic rhinitis.

SECONDARY OUTCOMES:
Total Nasal Symptom Score | 4 months
  To investigate the effect of repeat oral doses of ONO-4053 versus Cetirizine on nasal symptoms (Total Nasal Symptom Score) elicited by allergen chamber challenge in subjects with allergic rhinitis.
Total Ocular Symptom Score | 4 months
  Itching and ocular discharge monitored daily
Pharmacokinetics | Days 1 and 8
  AUE (0-2h, 2-6h and 0-6h)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Vienna Clinical Site, Vienna, Austria